CLINICAL TRIAL: NCT01196806
Title: Comparison of Measurement of Arterial Blood Pressure by L&T NIBP Module With Invasive Arterial Blood Pressure in Neonates
Status: Completed | Type: Observational
Sponsor: Larsen & Toubro Limited (Industry)
Responsible Party: L&T MEDICAL EQUIPMENT & SYSTEMS,MYSORE,INDIA, LARSEN & TOUBRO LIMITED
Other Study IDs: LTMED02-0910
Record Dates: First submitted 2010-09-06; First posted 2010-09-08 (Estimated); Last update posted 2010-09-08 (Estimated); Status verified 2010-09

CONDITIONS: Blood Pressure
Keywords: Non-Invasive Blood Pressure(NIBP)

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to compare Measurements of Arterial Blood Pressure by L&T NIBP Module With Invasive Arterial Blood Pressure in Neonates.

ELIGIBILITY:
Inclusion Criteria:

* Neonates admitted to NICU in whom arterial catheterization (radial or umbilical) was clinically indicated for a purpose other than for the comparative study.

Exclusion Criteria:

* All neonates in whom arterial catheterization was not clinically indicated.
* If minimum of 5-paired measurements is not obtained either due to technical or clinical reason.

Ages: 1 Minute to 30 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Total 20 numbers Neonates in NICU were studied during this study.
Sampling Method: Non-Probability Sample